CLINICAL TRIAL: NCT01105078
Title: Optimal Flow Rate During Cardiopulmonary Bypass
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Arndt-H. Kiessling, Head cardiovascular research, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI001AZ-AHK
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Tissue Perfusion
Keywords: cardiopulmonary bypass flow rate outcome tissue perfusion oxygenation l/min/m2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flow rate (Other): Comparison between a flow rate of 2.5/l/min/m2 versus 3.0/l/min/m2
  Interventions: Procedure: Flow rate

INTERVENTIONS:
Procedure: Flow rate — Different flow rate during cardiopulmonary bypass

SUMMARY:
Regardless of the development of cardiac surgery techniques and technologies, the question of an optimal extracorporeal circulation is still unanswered. There are globally accepted standards of perfusion, however, keep many of these procedures was not evidence-based review.

Generally accepted are flow rates during cardiopulmonary bypasses of 2.5 L/min/m2. This target was derived from the physiological conditions, but they are not the result of an adapted adjustment to the fundamentally non-physiological processes during extracorporeal circulation. Among other things, an increased metabolic demand during re-perfusion is not taken into account.

An increasing and optimizing of the standard flow rate of 0.5 L/min/m2 should be the aim of this investigation. Under optimal perfusion, the investigators are maintaining the microcirculation and organ protection in receipt of endothelial function and oxygen transport.

ELIGIBILITY:
Inclusion Criteria:

* Extracorporeal circulation
* Age > 18
* Written consent

Exclusion Criteria:

* Emergency cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-05; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Microcirulation | intraooperative
  measurement with O2C

CONTACTS AND LOCATIONS:
Locations (1):
- Johann Wolfgang Goethe University Hospital, Frankfurt am Main, Germany

REFERENCES:
- See also: Klinikum der Johann Wolfgang Goethe Universität Frankfurt aM Germany — http://www.kgu.de